CLINICAL TRIAL: NCT03650777
Title: Impact of Telehealth Warfarin Education on Patient Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 015-284
Record Dates: First submitted 2018-08-06; First posted 2018-08-29 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Educational Problems; Medication Adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Educational Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Warfarin Telehealth Education — Patients received education on warfarin through a video on an iPad, and were assessed on knowledge pre and post video, and at follow up visit

SUMMARY:
The objective of this study is to evaluate the effectiveness of telehealth warfarin education in a charity outpatient clinic. The purpose is to increase patient knowledge with regard to their warfarin therapy and to measure knowledge retention

DETAILED DESCRIPTION:
2. This study is conducted in outpatient ambulatory care clinics at the Baylor Family Medicine Worth Street clinic and the Irving Interfaith clinic. The average census for warfarin patients Friday clinic is 10. The anticoagulation clinic consists of an interdisciplinary team including physicians, medical assistants, nurse practitioners, and pharmacists. Patients initially visit with the provider and subsequent follow up INR checks are performed by the pharmacists or medical assistants. Currently, pharmacists manage the anticoagulation clinic on Fridays and medical assistants manage the clinic on Monday through Thursday. All providers provide patient education through written brochures.

3. Study Design

a. This study is a prospective, single-centered, randomized controlled quality improvement pilot study.

4. Warfarin Education Procedures

1. Each Friday morning, the pharmacist will identify the patients with appointments for INR checks.
2. As each patient checks in for their appointment, the pharmacist will ask the patient for consent to be a part of the study
3. If the patient says yes, the pharmacist will have the patient complete a warfarin questionnaire and health literacy test to see the patient's baseline knowledge on their warfarin therapy
4. Intervention patients (iPAD® video)

   1. The patient will then watch a warfarin education video on the iPAD®
   2. After the video the patient will receive point of care INR check and have their warfarin dose adjusted
   3. Patient will then complete the same warfarin questionnaire
   4. After completion, answers to the questionnaire will be presented to the patient. A written brochure will be given.
   5. A satisfaction survey will be given
   6. 30-60 days days later the pharmacist will follow up with the patient to repeat the warfarin questionnaire

   5. Description of iPAD video

a. Setting: a pharmacy b. Description: A pharmacist will provide education about warfarin using not only verbal instructions but also provide illustrations of directions. Please refer to Appendix for dialogue.

6. Control group

a. Patients' INR will be taken and warfarin education will be given verbally similar to Monday-Thursday clinic. A written brochure will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. English as a first language
3. Currently taking warfarin for an approved indication
4. Having the ability to see, read, and hear for verbal, written, and iPad® warfarin education

Exclusion Criteria:

1. Age < 18 years
2. Unwilling to receive iPad counseling
3. Cognitive dysfunction and impairments that prevents patient from fully comprehending warfarin education

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Knowledge Retention of Warfarin Education post video watching | pre and post video test(20 minutes)
  Difference in pre warfarin education video and post video test for warfarin education in patients receiving warfarin education via iPad
Long Term Knowledge Retention of warfarin education post video watching | initial and follow up visit (max 30 days)
  Difference in pre video test and follow up retention test for warfarin education in patients receiving warfarin education via iPad

SECONDARY OUTCOMES:
Self Reported Adherence to Warfarin therapy during duration of study | Between initial and follow up visit ( max 30 days)
  Descriptive results of patient self reported adherence (yes/no response) related to warfarin between initial and follow up visit
Satisfaction Survey | Max 30 days
  A satisfaction survey (designed by pharmacy resident) with 4 questions based on Likert scale (0-5), and one free response question patient completes on follow up visit. Name of Scale used for 4 questions: Likert. (Range 1-5, 1= highly disagree, 2= disagree, 3-neutral, 4-agree, 5-highly agree). There was no total of scoring, each response was individual of each other.
Adverse Events | Between initial and follow up visit ( max 30 days)
  Descriptive results of patient self reported adverse events related to warfarin between initial and follow up visit
Time of Warfarin in Therapeutic Range for Duration of Study | Between initial and follow up visit ( max 30 days)
  Time patient was within therapeutic range for their INR goal between initial and follow up visit

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heinrich K, Sanchez K, Hui C, Talabi K, Perry M, Qin H, Nguyen H, Tatachar A. Impact of an electronic medium delivery of warfarin education in a low income, minority outpatient population: a pilot intervention study. BMC Public Health. 2019 Aug 5;19(1):1050. doi: 10.1186/s12889-019-7370-4. PMID 31382942